CLINICAL TRIAL: NCT06491641
Title: The Effect of Nursing Care Based on Kolcaba's Comfort Theory on Comfort, Pain and Hemodynamic Variables of Babies in Neonatal Intensive Care Unit
Brief Title: The Effect of Nursing Care Based on Kolcaba's Comfort Theory on the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Fahri AŞKAN, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Fahri Aşkan
Record Dates: First submitted 2024-06-26; First posted 2024-07-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pain; Comfort Theory; Hemodynamic Variables
Keywords: pain; Comfort; Hemodynamic Variables; Kolcaba's Comfort Theory
MeSH Terms: conditions — Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental, randomised controlled, single-blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): During the application process, the babies in the experimental group will receive care based on Kolcaba's comfort theory during their stay in intensive care.
  Interventions: Other: Care based on Kolcaba's comfort theory
- Control Group (No Intervention): In this study, the control group will receive standard care.

INTERVENTIONS:
Other: Care based on Kolcaba's comfort theory — During the application process, the babies in the experimental group will receive care based on Kolcaba's comfort theory during their stay in intensive care.
  Other Names: Control Group
  Arms: Experimental Group

SUMMARY:
It was planned to determine the effect of nursing care based on Kolcaba's Comfort Theory on newborns' comfort, pain and hemodynamic variables for babies admitted to the neonatal intensive care unit.

* Does nursing care based on comfort theory reduce the comfort and pain levels of newborn babies?
* Does nursing care based on comfort theory have an effect on babies' vital signs?

DETAILED DESCRIPTION:
Comfort is defined as "an expected result with a complex structure within the physical, psychological, social and environmental integrity of helping the individual with his/her needs, providing peace of mind and being able to overcome problems." In his theory, Kolcaba defined comfort as "an expected result with a complex structure within the physical, psychospiritual, social and environmental integrity of helping the individual with his needs, providing peace of mind and overcoming problems."

The concept of comfort has been frequently used in neonatal intensive care units (NICU) and newborn babies in recent years. Unlike intrauterine life, NICU is an environment for newborn babies where there is noisy, cool, bright, dry, heat and light conditions are not good, and the baby has difficulty in making movements due to the power of gravity.

The physical structure of intensive care units (NICU), the anatomical and physiological immaturity of newborn babies, frequent routine care and invasive procedures may cause babies to lose their comfort.

This situation affects recovery and discharge times. Studies indicate that comfort is one of the most important factors affecting the speed of recovery.

The sample size of the study was determined using power analysis. The power of the research is defined as the possibility of revealing the difference between two applications. A study must have at least 80% power. It was calculated using the G. Power-3.1.9.4 program at the study's reliability coefficient of α=0.05 and 85% confidence level. In their study titled "The effect of the comfort care model on distress, pain and hemodynamic parameters in infants after congenital heart defect surgery", they found the effect size to be 0.816 and the minimum sample size to be 0.816. intervention with a theoretical power of 0.85. A total of 56 individuals will be included, 28 in the control group and 28 in the control group. Considering data loss, the study will be conducted with a total of 60 newborns, 30 newborns in each group.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with suspected or diagnosed sepsis
* Avoiding the use of analgesic, sedative or muscle relaxant drugs that may affect comfort.
* No congenital anomalies,
* Birth weight over 1500 grams,
* No need for mechanical ventilation,
* Vital signs are stable,
* Hospitalization of babies in the first 48 hours after birth,
* Newborn babies whose babies are deemed stable by the neonatologist will be included in the study.
* No hyperbilirubinemia requiring exchange transfusion,
* Those who do not have intrauterine infection (rubella, syphilis, toxoplasma) will be included in the study.

Exclusion Criteria:

* Newborns with sepsis or suspected sepsis
* Analgesic, sedative or muscle relaxant medication that may affect comfort is given,
* Enteral-fed infants,
* Having a congenital anomaly,
* Birth weight below 1500 grams,
* Those who require mechanical ventilation,
* Vital signs are unstable,
* Babies who are not hospitalized in the first 48 hours after birth,
* Newborn babies whose babies are not deemed stable by the neonatologist will not be included in the study.
* Those with hyperbilirubinemia requiring exchange transfusion,
* Those with intrauterine infection (rubella, syphilis, toxoplasma) will not be included in the study.

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale-Nips | It will be filled at the 0th hour of admission and then at the 24th, 48th and 72nd hour.
  The scale developed by Lawrence et al. is used for premature and newborns. In the neonatal pain scale, 5 (five) behavioral groupings (facial expression, crying, movements of arms and legs, state of wakefulness) and a physiological parameter (respiratory pattern) are evaluated and measured. Total score varies between 0-7. A high score on this scale indicates that the intensity of the pain is high. .
Newborn Comfort Behavior Scale | It will be filled at the 0th hour of admission and then at the 24th, 48th and 72nd hour.
  It is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. M. Each item in the scale is scored from 1 to 5. It is evaluated based on the total score. The lowest score that can be obtained from the Newborn Comfort Behavior Scale (YKDS) is 6 and the highest score is 30. If the total score of the scale is between 14-30, it is emphasized that the baby is in pain or distress, is uncomfortable and needs interventions to provide comfort. Scoring 4-6 on the Numerical Rating Scales indicates moderate pain and distress, while scoring 7-10 indicates severe pain and distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Tatvan Devlet Hastanesi, Bitlis, tATATVAN/BİTLİS, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided